CLINICAL TRIAL: NCT06365333
Title: Pneumatic Reduction For Intussusception In Children: A Retrospective Cohort Study In An Ultrahigh Volume Center
Brief Title: Pneumatic Reduction For Intussusception In Children: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Pediatric Surgeon, National Children's Hospital, Vietnam
Other Study IDs: 1451_04/BVNTW-VNCSKTE
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Intussusception
Keywords: Intussusception; Minimally invasive; Laparoscopic; Pediatric; Air enema; Pneumatic reduction
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FGAR-treated: Patients diagnosed with idiopathic intussusception, admitted to the National Children's Hospital between January 2016 and December 2017, exhibiting clinical signs and symptoms consistent with intussusception, and confirmed via ultrasound examination
  Interventions: Procedure: Fluoroscopic-guided air-enema reduction (FGAR)

INTERVENTIONS:
Procedure: Fluoroscopic-guided air-enema reduction (FGAR) — A hand-held pump facilitated the delivery of atmospheric air, while pressure was monitored using a digital gauge. A two-way Foley's balloon catheter, ranging from 18oF to 24oF in diameter depending on age, was inserted rectally to introduce air. Following insertion, the balloon was filled with 10cc of saline to prevent air leakage, with patient immobilization ensured by leg straps and hand positioning above the head for abdominal exposure. Under intermittent fluoroscopy, the surgeon operated the pump with the right hand, inflating the catheter to 80 to 120 mmHg, simultaneously palpating the intussusceptum with the left hand, employing a deep gliding motion for deep and fixed cases. Successful reduction, indicated by air entry into the small bowel, was confirmed under fluoroscopy, with a subsequent brief rotating abdominal massage ensuring uniform air distribution throughout the small intestine, confirming complete reduction.

SUMMARY:
In pediatric patients, intussusception predominantly occurs in the ileocecal region, with over 90% of cases lacking identifiable causative factors, initiating through peristalsis-driven invagination of bowel segments leading to compromised blood flow and subsequent bowel edema. Persistent obstruction may progress to bowel ischemia and infarction. Vietnam exhibits a higher incidence of intussusception compared to other countries, albeit with similar clinical presentations and anatomical locations, hinting at shared pathophysiology. Despite evidence supporting the safety and efficacy of non-surgical reduction techniques, many medical centers in low- to middle-income countries (LMICs) have not adopted these methods, resulting in unnecessary surgical interventions. The Vietnam National Hospital of Pediatrics (NCH) has employed air enema reduction since the early 2000s but lacks a comprehensive study on fluoroscopic-guided air-enema reduction (FGAR) techniques or success rates. Thus, this study aims to evaluate the long-term outcomes of pneumatic reduction for intussusception at NCH, a high-volume institution in a lower-middle-income country.

DETAILED DESCRIPTION:
In pediatric patients, intussusception primarily occurs in the ileocecal region, with more than 90% of cases lacking identifiable causative factors. The invagination of bowel segments is propelled by peristalsis, leading to compromised blood flow. This venous occlusion precipitates bowel edema, and if the obstruction persists, it can progress to bowel ischemia and infarction. The incidence of intussusception in Vietnam exceeds that of any other country with available data on incidence rates. Despite variations in incidence rates, intussusception's clinical presentation and anatomical location remain largely consistent between Vietnam and other countries, suggesting a common underlying pathophysiology. Many medical centers in low- to middle-income countries (LMICs) have yet to adopt these non-surgical approaches, resulting in unnecessary surgical interventions for a significant portion of patients. At the Vietnam National Hospital of Pediatrics (NCH), air enema reduction has been a standard practice since the early 2000s. Nonetheless, there has been no comprehensive study delineating the technique of fluoroscopic-guided air-enema reduction (FGAR) at NCH, nor assessing its success rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with idiopathic intussusception, admitted to the National Children's Hospital between January 2016 and December 2017, exhibiting clinical signs and symptoms consistent with intussusception, and confirmed via ultrasound examination.
* Fluoroscopy-guided pneumatic reduction was performed with a maximum of three attempts. Patients who did not respond to pneumatic reduction underwent minimally invasive surgical intervention, either laparoscopic reduction or trans-umbilical mini-open reduction.

Exclusion Criteria:

* Patients demonstrating clinical instability characterized by signs of peritonitis or intestinal perforation necessitating conventional laparotomy.
* Patients deemed unsuitable for air enema reduction due to a grossly distended abdomen or compromised cardiopulmonary function.

Ages: 2 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients diagnosed with idiopathic intussusception admitted to the National Children's Hospital between January 2016 and December 2017
Sampling Method: Non-Probability Sample
Enrollment: 3562 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Complicated intussusception | through study completion (2 years)
  Complications, including bowel perforation, occurred during FGAR
ICU admission | through study completion (2 years)
  Clinically unstable patients post-FGAR that required ICU admission
Death | through study completion (2 years)
  Mortality or severe morbidity noted post-FGAR
Failed FGAR | through study completion (2 years)
  Unsuccessful reduction that requires transition to surgical intervention
Recurrence | through study completion (2 years)
  Recurrence of intussusception during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (2):
- Vietnam (2):
  - The National Hospital of Pediatrics, Hanoi
  - Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bines JE, Liem NT, Justice FA, Son TN, Kirkwood CD, de Campo M, Barnett P, Bishop RF, Robins-Browne R, Carlin JB; Intussusception Study Group. Risk factors for intussusception in infants in Vietnam and Australia: adenovirus implicated, but not rotavirus. J Pediatr. 2006 Oct;149(4):452-60. doi: 10.1016/j.jpeds.2006.04.010. PMID 17011313
- [Background] Tran LA, Yoshida LM, Nakagomi T, Gauchan P, Ariyoshi K, Anh DD, Nakagomi O, Thiem VD. A High Incidence of Intussusception Revealed by a Retrospective Hospital-Based Study in Nha Trang, Vietnam between 2009 and 2011. Trop Med Health. 2013 Sep;41(3):121-7. doi: 10.2149/tmh.2013-09. Epub 2013 Aug 20. PMID 24155653
- [Background] Chowdhury TK, Ahsan MQ, Chowdhury MZ, Chowdhury MTS, Imam MS, Alam MA, Farooq MAA. Hydrostatic reduction of intussusception with intermittent radiography: an alternative to fluoroscopy or ultrasound-guided reduction in low-income and middle-income countries. World J Pediatr Surg. 2021 Jan 14;4(1):e000221. doi: 10.1136/wjps-2020-000221. eCollection 2021. PMID 36474637
- [Background] Trang NV, Burnett E, Ly LH, Anh NP, Hung PH, Linh HM, Trang NCT, Canh TM, Minh VT, Tate JE, Yen C, Anh DD, Parashar UD. Recurrent intussusception among infants less than 2 years of age in Vietnam. Vaccine. 2018 Dec 14;36(51):7901-7905. doi: 10.1016/j.vaccine.2018.02.056. Epub 2018 Feb 23. PMID 29478753
- [Background] Hailemariam T, Sisay S, Mebratu Y, Belay F, Getinet T, Solomon S, Belina M, Abebe A, Hilawi Tewodros B, Manyazewal T. Effects of sedatives on radiologic enema reduction in children with ileocolic intussusception: A systematic review and meta-analysis. Eur J Radiol. 2024 Jan;170:111237. doi: 10.1016/j.ejrad.2023.111237. Epub 2023 Nov 27. PMID 38039783
- [Background] Khorana J, Tepjuk S, Singhavejsakul J, Tepmalai K, Chantakhow S, Ukarapol N, Damrongmanee A, Samerchua A, Bunchungmongkol N, Visrutaratna P, Morakote W, Nate-Anong B, Chanaturakarnnon S, Itthidecharon K, Chaimongkhon P. A comparison of the success rate of pneumatic reduction in intussusception between general anesthesia and deep sedation: a randomized controlled trial. Pediatr Surg Int. 2023 Apr 25;39(1):186. doi: 10.1007/s00383-023-05474-2. PMID 37095299
- [Background] Xie X, Wu Y, Wang Q, Zhao Y, Chen G, Xiang B. A randomized trial of pneumatic reduction versus hydrostatic reduction for intussusception in pediatric patients. J Pediatr Surg. 2018 Aug;53(8):1464-1468. doi: 10.1016/j.jpedsurg.2017.08.005. Epub 2017 Aug 8. PMID 28827051
- [Background] Beres AL, Baird R. An institutional analysis and systematic review with meta-analysis of pneumatic versus hydrostatic reduction for pediatric intussusception. Surgery. 2013 Aug;154(2):328-34. doi: 10.1016/j.surg.2013.04.036. PMID 23889959
- [Background] Chew R, Ditchfield M, Paul E, Goergen SK. Comparison of safety and efficacy of image-guided enema reduction techniques for paediatric intussusception: A review of the literature. J Med Imaging Radiat Oncol. 2017 Dec;61(6):711-717. doi: 10.1111/1754-9485.12601. Epub 2017 Apr 17. PMID 28419712
- [Background] Okumus M, Emektar A. Pediatric intussusception and early discharge after pneumatic reduction. Acta Chir Belg. 2019 Jun;119(3):162-165. doi: 10.1080/00015458.2018.1487190. Epub 2018 Jun 27. PMID 29947299
- [Background] Cox S, Withers A, Arnold M, Chitnis M, de Vos C, Kirsten M, le Grange SM, Loveland J, Machaea S, Maharaj A, Madhi SA, Tate JE, Parashar UD, Groome MJ. Clinical presentation and management of childhood intussusception in South Africa. Pediatr Surg Int. 2021 Oct;37(10):1361-1370. doi: 10.1007/s00383-021-04946-7. Epub 2021 Jul 2. PMID 34213589
- [Background] Wong CW, Chan IH, Chung PH, Lan LC, Lam WW, Wong KK, Tam PK. Childhood intussusception: 17-year experience at a tertiary referral centre in Hong Kong. Hong Kong Med J. 2015 Dec;21(6):518-23. doi: 10.12809/hkmj144456. Epub 2015 Sep 11. PMID 26371157
- [Background] Burnett E, Kabir F, Van Trang N, Rayamajhi A, Satter SM, Liu J, Yousafzai MT, Anh DD, Basnet AT, Flora MS, Houpt E, Qazi SH, Canh TM, Rayamajhi AK, Saha BK, Saddal NS, Muneer S, Hung PH, Islam T, Ali SA, Tate JE, Yen C, Parashar UD. Infectious Etiologies of Intussusception Among Children <2 Years Old in 4 Asian Countries. J Infect Dis. 2020 Apr 7;221(9):1499-1505. doi: 10.1093/infdis/jiz621. PMID 31754717
- [Result] Yang H, Wang G, Ding Y, Li Y, Sun B, Yue M, Wang J, Song D. Effectiveness and safety of ultrasound-guided hydrostatic reduction for children with acute intussusception. Sci Prog. 2021 Jul-Sep;104(3):368504211040911. doi: 10.1177/00368504211040911. PMID 34519571
- [Result] Wang Z, He QM, Zhang H, Zhong W, Xiao WQ, Lu LW, Yu JK, Xia HM. Intussusception patients older than 1 year tend to have early recurrence after pneumatic enema reduction. Pediatr Surg Int. 2015 Sep;31(9):855-8. doi: 10.1007/s00383-015-3726-8. Epub 2015 Jul 14. PMID 26169529
- [Result] Khorana J, Singhavejsakul J, Ukarapol N, Laohapensang M, Wakhanrittee J, Patumanond J. Enema reduction of intussusception: the success rate of hydrostatic and pneumatic reduction. Ther Clin Risk Manag. 2015 Dec 15;11:1837-42. doi: 10.2147/TCRM.S92169. eCollection 2015. PMID 26719697
- [Result] Elzeneini WMA, Cusick E. A large single-center experience in management of pediatric intussusception. Pediatr Int. 2023 Jan-Dec;65(1):e15495. doi: 10.1111/ped.15495. PMID 36749147
- [Result] Delgado-Miguel C, Garcia A, Delgado B, Munoz-Serrano AJ, Miguel-Ferrero M, Barrena S, Lopez-Santamaria M, Martinez L. Intussusception Management in Children: A 15-Year Experience in a Referral Center. Indian J Pediatr. 2023 Dec;90(12):1198-1203. doi: 10.1007/s12098-022-04248-3. Epub 2022 Jul 12. PMID 35821554
- [Result] Younes A, Lee S, Lee JI, Seo JM, Jung SM. Factors Associated with Failure of Pneumatic Reduction in Children with Ileocolic Intussusception. Children (Basel). 2021 Feb 12;8(2):136. doi: 10.3390/children8020136. PMID 33673183
- [Result] Carapinha C, Truter M, Bentley A, Welthagen A, Loveland J. Factors determining clinical outcomes in intussusception in the developing world: Experience from Johannesburg, South Africa. S Afr Med J. 2016 Jan 12;106(2):177-80. doi: 10.7196/SAMJ.2016.v106i2.9672. PMID 26821898